CLINICAL TRIAL: NCT01213329
Title: Immunophenotyping and Functional Profiles of Peripheral Lymphocytes in Renal Transplant Recipients After T-cell Depletion With Alemtuzumab (Anti-CD52 Monoclonal Antibody)-Potential Implications for Safe Immunosuppressive Minimization
Brief Title: Immunophenotyping of Peripheral T Cells After T Cell Depletion With Alemtuzumab
Status: Terminated | Phase: Phase 4 | Type: Interventional
Sponsor: Northwestern University (Other)
Collaborators: American Society of Transplant Surgeons (Other)
Responsible Party: Principal Investigator, Lorenzo Gallon, Associate Professor of Medicine & Surgery, Northwestern University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STU00011048
Record Dates: First submitted 2010-09-30; First posted 2010-10-04 (Estimated); Results first posted 2011-07-04 (Estimated); Last update posted 2019-04-10 (Actual); Status verified 2019-03

CONDITIONS: Kidney Transplant
MeSH Terms: interventions — Alemtuzumab

STUDY DESIGN:
Intervention Model Description: Phase 1: 50 subjects were to receive study intervention. If any subjects demonstrated persistent donor specific unresponsiveness at the 12 month post-transplant time point, they would proceed into Phase 2. In that phase, the unresponsive subjects would have been randomized to one of three arms that would modify their standard of care immunosuppression.
  None of the 50 subjects from Phase 1 demonstrated persistent donor specific unresponsiveness, therefore, phase 2 was never started.
Oversight: Data Monitoring Committee: No

ARMS (1):
- Phase I: Alemtuzumab (Experimental): During Phase I Portion: Each kidney transplant recipient received one 30mg dose (IV push)of Alemtuzmab in the operating room per Standard of Care.
  Interventions: Drug: Alemtuzumab

INTERVENTIONS:
Drug: Alemtuzumab — All kidney transplant recipients received one 30mg dose (IV push) of Alemtuzumab in operating room per Standard of Care.
  Other Names: Campath 1-H®

SUMMARY:
The purpose of this study is to check the T and B cells of the immune system in 50 newly transplanted patients whom have received a kidney (50 recipients and 50 donors totaling 100 anticipated participants). This will be done to see how the Standard of Care (SOC) anti-rejection medication, Alemtuzumab (Campath 1-H®) affects these cells- Campath 1-H® reduces the number of T cells produced by one's body.

DETAILED DESCRIPTION:
The purpose of this study is to check the T and B cells of the immune system in 50 newly transplanted patients whom have received a kidney (50 recipients and 50 donors totaling 100 anticipated participants). This will be done to see how the Standard of Care (SOC) anti-rejection medication, Alemtuzumab (Campath 1-H®) affects these cells- Campath 1-H® reduces the number of T cells produced by one's body. We will look for these cells using a number of laboratory tests; It will require the subjects to each give 65mL of blood at each of the 3 visits that occur during phase 1. Up to 12 subjects will be chosen from phase 1 to participate in phase 2 depending on lab results.

In phase 2, subjects will be randomized to one of the three following groups:

Group one: Continue normal immunosuppression with tacrolimus and Cellcept® (control group)

Group two: Cellcept® will be tapered down to 70% in three months. Tacrolimus will be continued at the same dosage.

Group three: Tacrolimus will be reduced to 70% in three months. Cellcept® will be continued at the same dosage.

There will be an analysis of these cells at different time point, pre and post kidney transplant. The data collection will allow us to study the stability over time of particular phenotypes (cell structures) and T cell function. We will also evaluate how the two different "minimizing protocols" effect the cell structure. Results from laboratory testing may allow us to define certain criteria that can be broadly applied in solid organ transplant recipients. This may allow for safe reduction of the anti-rejection medication that transplant recipients receive.

ELIGIBILITY:
Inclusion Criteria:

1. Adult subjects between ages 18-65 years old of either gender
2. Recipients have an available ABO compatible living donor for transplant
3. Subjects are listed to be a single-organ transplant recipient (kidney only)
4. Subjects have the ability to provide informed consent

Exclusion Criteria:

1. Subjects have panel reactive antibody greater than 35%
2. Subjects have the potential to have a high recurrence rate of their primary renal disease (i.e. Focal Segmental Glomerulonephritis )
3. Subjects who have a history of Hepatitis C
4. Subjects who have had a previous organ transplant
5. Subjects are unable to fully understand the purpose of the study, thereby unable to give a fully informed consent
6. Subjects with a positive lymphocytotoxic crossmatch using donor lymphocytes and recipient serum
7. Subjects who are pregnant or nursing
8. Subjects who, due to the existence of a surgical, medical or psychiatric condition, other than the current transplant, which in the opinion of the investigator, precludes enrollment into this trial.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2006-02; Primary Completion 2009-04 (Actual); Study Completion 2009-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lorenzo Gallon, MD, Principal Investigator — Northwestern University, Northwestern Memorial Hospital, Northwestern Medical Faculty Foundation
Locations (1):
- Northwestern Memorial Hospital, Chicago, Illinois, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: All patients were approached pre-operatively in the transplant clinic at Northwestern Memorial Hospital. Recruitment began on July 28, 2005 and lasted until April 14, 2008.
Pre-assignment Details: The first year of the study was specimen collection only. Group assignment (phase 2) was intended to begin after 12months of sample collection and there were not any subjects who continued into phase 2. An additional pair enrolled compared to the number that started this study. This is due to a loss of samples from a processing inconsistency
Groups:
- Alemtuzumab (Phase I): All transplant recipients received one 30mg dose (intravenous "IV" push)of Alemtuzmab in the operating room per Standard of Care.
Period: Screening
Arm/Group | Alemtuzumab (Phase I) | Donor Comparison
Started | 25 | 25
Completed | 25 | 25
Not Completed | 0 | 0
Period: Phase 2
Arm/Group | Alemtuzumab (Phase I) | Donor Comparison
Started | 0 (No subjects continued into phase 2.This is due to a loss of samples from a processing inconsistency.) | 0 (No subjects continued into phase 2.This is due to a loss of samples from a processing inconsistency.)
Completed | 0 | 0
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Alemtuzumab (Phase I) | Donor Comparison | Total
Number analyzed (Participants) | 26 | 25 | 51
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 26 | 25 | 51
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 41 (22) | 43 (9.46) | 42 (31.46)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 13 | 18
  Male | 21 | 12 | 33
Region of Enrollment [Number; unit: participants]
  United States | 26 | 25 | 51

OUTCOME MEASURES:

1. Primary Outcome: The Effect of T Cell Depletion on Phenotypic & Functional Profiles of Peripheral Blood Mononuclear Cells in Steroid-free Kidney Transplant Recipients.
Description: Blood was collected to assess peripheral blood leukocytes prior to kidney transplant, 6 months & 12 months post-transplant as follows: to obtain absolute count of circulating CD4, CD8 positive T cells, B cells & NK cells, naive & memory cells (CD45RA, CD45RO), activated T cells (CD4/CD38, CD8/CD38), regulatory cells (CD4+ CD25+). Unfortunately blood samples were lost due to malfunction of liquid nitrogen tank that stopped working during a power loss.
Time Frame: Pre-transplant, 6months & 12 months post-transplant
Population: samples from 26 recipient/donor pairs were collected = 52 collected but no analysis was performed because samples were lost.
Arm/Group | Alemtuzumab (Phase I)
Number analyzed (Participants) | 0

2. Secondary Outcome: Donor Specific Hypo-reactivity.
Description: Identify, by studying recipients for development of donor specific hypo-reactivity and through immunopathologic analysis of renal allograft biopsies, immunologically stable renal transplant patients in whom immunosuppression can be safely minimized.
  Unfortunately this secondary outcome was not studied because of lost samples that did not allowed us further analysis to identify patients with donor specific hypo reactivity.
Time Frame: Pre-transplant, 6mo & 12mo post-transplant
Population: no one were analyzed due to loss of blood samples
Groups:
- Donor Comparison: The donor group served as source of PBMCs to use as stimulator for the patients that received Alemtuzumab.
Arm/Group | Donor Comparison
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: The period in which adverse events data was collected began with the first day of enrollment and ended at the final study visit: February 2006 through April 2009.
Arm/Group | Alemtuzumab (Phase I) | Donor Comparison
Serious Adverse Events (participants affected / at risk) | 0/26 | 0/25
Other Adverse Events (participants affected / at risk) | 0/26 | 0/25

LIMITATIONS AND CAVEATS:
Processing of blood samples was inconsistent and lab results were questionable. Research blood specimens were in addition to Standard of Care (SOC) required blood. Most research visits were planned at the same time as SOC visits.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes